CLINICAL TRIAL: NCT06016647
Title: Precision Multi-Axis Pain Assessment of Injured Workers to Improve Treatment and Work Outcomes
Brief Title: Multi-axis Assessment of Injured Workers
Status: Recruiting | Type: Observational
Sponsor: Dave Walton (Other)
Collaborators: CBI Health (Unknown)
Responsible Party: Sponsor-Investigator, Dave Walton, Associate Professor, School of Physical Therapy (cross-appt. Dept. of Psychiatry), Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: 121883
Record Dates: First submitted 2023-08-16; First posted 2023-08-30 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Injury; Musculoskeletal Strain; Low Back Pain; Neck Pain; Upper Extremity Injury; Lower Extremity Problem; Work-related Injury
MeSH Terms: conditions — Low Back Pain; Neck Pain; Arm Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Musculoskeletal-specific WSIB programs of care — Clinicians within this network provide care under a standardized framework that limits confounding from different interventions and the researchers will not manipulate treatment decisions.

SUMMARY:
The percentage of loss time claims receiving Loss of Earnings benefits at 3 months has continued to rise amongst injured workers in Ontario despite the Workplace Safety and Insurance Board (WSIB) approach of "Better at Work". The primary health services to address loss time claims associated with musculoskeletal injuries include the evidenced-based programs of care, occupational health assessment program and musculoskeletal specialty programs, however, these are set to be revised and relaunched in Q1 2023. Across treatment protocols there are challenges that, at least in part, appear to contribute to the increasing percentage of workers on full loss of earnings at 3 months include (1) inconsistent early identification of workers who should be triaged to various health services and (2) reliable determination of the optimal timing of referral to the most targeted care to enable a safe and sustainable return to work. The investigators aim to develop and evaluate a predictive assessment model to triage workers to the best service within the first 8 weeks of their claim to increase the rate of early return to work, with the long-term goal that the triage protocol becomes part of a person-centric protocol that reduces the duration of work-related disability.

The investigators will develop and evaluate an assessment protocol for injured workers that enter any of the musculoskeletal-specific WSIB programs of care, which have been consolidated into a single program as of 2023. This study will be a prospective inception cohort design using data collected from injured workers receiving WSIB musculoskeletal programs of care services at CBI Health clinics in Ontario Canada. Worker data will be collected at intake to the program of care service and again approximately four and eight weeks after intake (or earlier if a worker completes the program of care). The investigators will complete data analysis in three steps including descriptive and bivariate associations, Maximum Likelihood-based Latent Profile Analysis, and evaluation of results against successful work outcomes and secondary outcomes. Qualitative data will be mined for alternative indicators of recovery / non-recovery. The study recruitment goal is 300 - 350 workers with complete follow-up within a 2-year period.

DETAILED DESCRIPTION:
Background and Rationale It has long been known that early and targeted acute-stage intervention is the best way to prevent chronic pain. For 15 years the Principal Investigator has been developing novel tools, strategies, and frameworks for predicting and preventing the acute-to-chronic transition in other populations. These include self-report tools that have individually demonstrated >75% accuracy in predicting 12-month outcomes when administered in the first weeks from injury, new interpretations of common pain assessment and evaluation tools, and new frameworks for understanding pain and its management at both the acute and chronic stages. The investigators have used advanced analytic techniques to identify and describe the recovery trajectories present in a sample of people with mixed musculoskeletal injuries using data collected within days to weeks, predicting outcomes up to 12 months post-injury. In a recently-completed project, some of these innovations were integrated into a single online questionnaire targeting Canadian military veterans with chronic pain. The results of that analysis revealed a 5-cluster solution based on responses to self-report measures of 7 domains (or axes) of drivers of the pain experience. The investigators believe this strategy will also have value when translated and implemented in more acutely injured workers in Canada as a single risk stratification and management protocol. The longer-term goal is to use this type of simple self-assessment protocol to empower injured workers and claims managers to triage into the right care pathway, reduce time off work, and improve the likelihood of successful outcomes.

Based on our team's extensive work in the prognosis of post-traumatic musculoskeletal injuries, the investigators propose that it is possible to identify those who can be expected to achieve a full return to work within only the programs of care and differentiate them from those who will experience some form of delayed or non-return to work and can do so within the first 3 weeks (21 days) from injury with >80% accuracy.

Objective Development and validation of a multi-axis 'risk/prognosis' worker-reported screening tool comprising tools that can be administered within the first 8 weeks of work-related injury and provide >80% accuracy in predicting work recovery trajectories over the subsequent 2 months.

Recruitment Recruitment will occur through CBIH programs of care provider clinics for injured workers, using both emailed and posted invitations. In both cases explicit opt-in consent will be obtained for this study following the protocol for digital online consent procedures from Western's Research Ethics Board (REB).

Members of the research team at Western will monitor the portal for new participants daily. New participants will be entered into a Master List that includes only name, contact email address, and a study-specific randomly-generated 4-digit ID number. The Master List is necessary to permit the linking of responses across data collection periods and will be stored separately from the raw data file that will include only ID number. The research team member will subsequently create a unique survey link tied to the participant's email addresses and send that to the participant within two working days. That survey will start with the screening questions for inclusion. Those who pass the screen will proceed with the full set of survey questions, while those who are screen-failed will be presented with a thank participant screen and their study involvement will end. Upon entry into the Master List, follow-up dates at 1 and 2 months post-inception will be automatically calculated, and the research team members will use those to ensure follow-up survey forms are sent on time.

Clinician Feedback: The emailed link to the clinician feedback survey will be sent to all members of the CBI Health Inc. network of physiotherapists in Canada, along with the new classification tool/algorithm. The CBI Health collaborators on this protocol will facilitate dissemination of the link through internal CBI Health email channels. Any clinician who is a registered physiotherapist within the CBI Health Inc. network will be eligible to participate. They will receive the new stratification algorithm and a link to a single-page feedback survey. In this way emails will be stored in a separate database from survey responses. The list of emails will remain with the Western researchers and will not be shared with the CBI Health leadership.

Methodology This is an observational prospective inception cohort using data collected from injured workers entering one of the CBIH programs of care. Clinicians within this network provide care under a standardized framework that limits confounding from different interventions and the researchers will not manipulate treatment decisions.

Duration: All eligible Workers will be invited to participate. Participants will be in the study for two months (8 weeks) total, from inception to outcome. A single interim data collection at 4 weeks post-inception will permit longitudinal trajectories to be established for each outcome as a tertiary analytic target (interpreted as slope/rate of recovery).

DATA ANALYSIS: 1. Descriptive and bivariate associations to describe the sample and evaluate associations between the predictors and the outcomes; 2. Maximum likelihood-based latent profile analysis in which the predictors (and their subscales where available) are used to identify meaningful profiles ('clusters') of injured Workers. This will be guided by 3 core principles of i) statistical justification, ii) parsimony, and iii) clinical meaningfulness; 3. The profiles will then be evaluated to determine the proportion of successful primary (work) and secondary outcomes within each. The investigators anticipate that one profile will comprise a majority who achieve Full return to work by 8 weeks and another will comprise a majority who fail to achieve return to work, with other clusters including mixed outcomes. Prognostic accuracy of the new clusters will also be compared against the TIDS to determine whether the use of additional scales offers improved utility over the single scale.

SAMPLE SIZE: Prior authors have endorsed at least 250 unique people in the data for robust Maximum likelihood-based latent profile analyses, and our own work in a sample of Canadian military veterans with chronic pain that used almost identical indicators to the current project successfully identified 5 latent classes with n = 322 respondents. The investigators will target up to n = 350 over a two-year project window.

Quality Assurance: All Western members of the research team have completed either or both of the Good Clinical Practice or Tri-Council Policy Statement 2 training modules. Certificates of completion are available upon request. Further, the Principal Investigator has completed the CIHR Institute of Gender training module on sex- and gender-based analyses, Equity, Diversity and Inclusion training through Western University, and Ownership, Control, Access and Possession training for research with Indigenous peoples.

The investigators acknowledge a potential for conflict of interest regarding the collaboration with the CBIH team. Importantly, CBIH will be instrumental for helping meet the recruitment targets as one of Canada's largest networks of rehabilitation providers for injured workers. Members of the CBIH team will also be critical for ensuring the design described herein can be expected to lead to implementable findings, and they will facilitate clinical interpretation of analytic results, and facilitate dissemination of the findings throughout their network of clinics. Importantly, all findings of this work will be published in scientifically-rigourous peer-reviewed journals relevant to the field, and no part of the data or findings will be the proprietary property of CBIH. Participants will be made aware of this arrangement prior to providing their informed consent to participate.

Expected Outcomes:

This work is anticipated to result in a new risk/prognosis screening tool to discriminate between those injured workers most likely to transition back to full return to work quickly from those most likely to experience delayed or incomplete recovery, and the investigators further anticipate that the latent classes identified will be useful for directing injured workers to the most appropriate health discipline in the patient-centred spirit of 'right care, right person, right time'. Logical next steps from this work will be to use the most accurate predictor variables found herein to create and test intervention strategies that specifically target the risks present in higher-risk injured workers. Through this program of research, the investigators anticipate reducing the burden of delayed return to work borne by both injured workers and those who insure them.

Ethics: All methods for this study have been approved by the Health Sciences Research Ethics Board of Western University (London Ontario, Canada), REB No. 121883, having been evaluated by an independent peer reviewer against the standards of the Declaration of Helsinki and in accordance with the Tri-Council Policy Statement 2.

ELIGIBILITY:
Inclusion Criteria: Eligible participants are those aged ≥18 years, able to read 6th grade English, presenting to a program of care for rehabilitation of a workplace injury with a primary musculoskeletal or Low Back Pain component.

Exclusion Criteria: Participants with significant cognitive impairment or learning disability (self-reported) that interfere with following multi-step instructions will be excluded from this study. The exclusive focus on those entering program of care-based rehab will naturally exclude workers with catastrophic injuries (e.g., loss of limb, multiple fractures, burns) or those for whom a mental health disorder (e.g., PTSD, depression) is the primary diagnosis, thereby homogenizing the types of injuries included.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective inception cohort using data collected from injured workers entering one of the CBIH programs of care.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Work status | 8 weeks
  Full Return-to-Work, Return-to-Work with temporary restrictions, or redirected to other treatment options. With the Full RTW category serving as the reference against which the other outcomes will be considered.

SECONDARY OUTCOMES:
Pain severity | 8 weeks
  Brief Pain Inventory: These are four 0-10 rating scales that ask about pain at its best, least, on average, and right now. Reported as a mean out of 10 where a higher score indicates more intense pain.
EuroQoL-5D (EQ5D-5L) | 8 weeks
  EuroQoL-5D and the three additional questions. The EQ-5D has been used in its original form, and we have added 3 additional questions related to fatigue, sleep, and connections with others that patient partners have repeatedly indicated are important but are not captured in the current scale. For purposes of this analysis, and in keeping with terms of use of the EQ-5D-5L, those final 3 questions will be interpreted separately from the original items for reporting purposes. A final question on how the respondent has defined their sense of recovered/not recovered will be collected through open text to give richer information on the ways that injured workers make sense of the very notion of what it is to be 'recovered' from a workplace injury. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
Body diagram | 8 weeks
  An interactive 'body diagram', or pain map, will be provided to allow participants to indicate the areas and extent (distribution) of their pain, which will be evaluated as a secondary prognostic indicator under the hypothesis that more widespread pain is a poor prognostic indicator for rapid recovery. Reported as a total number of shaded areas, where a higher number represents more widespread pain.

OTHER OUTCOMES:
MultiDimensional Symptom Index (MSI) | 8 weeks
  The MultiDimensional Symptom Index (MSI), a 10-item self-report tool that uses a scoring matrix to create a profile of symptom type, frequency, and interference across 10 different symptom types. It will be primarily used to discriminate between pain of nociceptive (primarily somatic) origin (scale range 0-50) and that of more central (non-somatic) dominance (scale range 0-62). A higher score on either subscale represents a worse pain state.
A shortened 4-item version of The Self-Report version of the Leeds Assessment of Neuropathic Signs and Symptoms (S-LANSS). | 8 weeks
  A shortened 4-item version of The Self-Report version of the Leeds Assessment of Neuropathic Signs and Symptoms (S-LANSS). The S-LANSS is a 7-item scale with each item offering a simple yes/no response option. It has been well-validated against clinical diagnoses of neuropathic pain with a score ≥12 providing over 80% accuracy. We have previously used statistical triangulation to identify 4 of the items that combined provide a nearly perfect association with the full 7 items and offers the advantage of brevity.
The Fremantle Body Awareness questionnaire - general version (FreBAQ-general) | 8 weeks
  The Fremantle Body Awareness questionnaire - general version (FreBAQ-general). This is a 6-item questionnaire (range 0-24) derived from original version of the FreBAQ, dedicated to specific body regions (e.g., back, neck, knee, shoulder) that makes use of digital text piping to first ask the respondent about their most problematic body region, then uses that answer to populate the 6 FreBAQ-general items. A higher score indicates a greater sense of sensorimotor disconnection with painful body regions.
The Brief Pain Catastrophizing Scale (BriefPCS-4) | 8 weeks
  The Brief Pain Catastrophizing Scale (BriefPCS-4), a 4-item version of the original 13-item PCS that captures catastrophic beliefs about pain, such as 'it's awful and I feel that it overwhelms me'. The 4 items were correlated with the full 13-item version at r = 0.97 in a prior study, providing a near-perfect estimate of the full version with lower respondent burden. The scale range is 0-16 with a higher number indicating more catastrophic beliefs about pain.
The short Patient Health Questionnaire-4 item version | 8 weeks
  The short Patient Health Questionnaire-4 item version. This tool comprises two items useful as a brief screen for anxiety disorders and two as a brief screen for depressive disorders. With so few items it is far more sensitive than specific as a diagnostic tool, but as a combined score it provides a metric of negative emotional state on a 0-12 scale where a higher number represents greater emotional distress.
The Intersectional Discrimination Index - Major (InDI-M) | 8 weeks
  The Intersectional Discrimination Index - Major (InDI-M), a newer 13-item questionnaire is intended to capture experiences of discrimination/exclusion or interpersonal violence perpetrated against the respondent that is perceived to have been due to some aspect of their identity (e.g., skin colour, sex, gender, body size, age, disability, etc…). We have previously used this tool in a sample of military veterans with chronic pain and found that it shows a small but significant association with pain severity, and is a dominant driver in one sub-category of that sample with a trauma-dominant pain profile. Scale range is 0-26 with a higher score indicating more experiences of intersectional discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: David Walton, PhD, Principal Investigator — CANSpine Lab, School of Physical Therapy, Western University, Canada
Locations (1):
- CBI Health, Multiple Locations, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, we will pursue options for making the de-identified data open-access through engagement with the REB around safe and ethical data sharing.
Supporting Information: Analytic Code
Time Frame: Upon study completion
Access Criteria: Open access and administrative database.

REFERENCES:
- [Background] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Tein JY, Coxe S, Cham H. Statistical Power to Detect the Correct Number of Classes in Latent Profile Analysis. Struct Equ Modeling. 2013 Oct 1;20(4):640-657. doi: 10.1080/10705511.2013.824781. PMID 24489457
- [Background] Lee JY, Walton DM, Tremblay P, May C, Millard W, Elliott JM, MacDermid JC. Defining pain and interference recovery trajectories after acute non-catastrophic musculoskeletal trauma through growth mixture modeling. BMC Musculoskelet Disord. 2020 Sep 17;21(1):615. doi: 10.1186/s12891-020-03621-7. PMID 32943021
- [Background] Modarresi S, Suh N, Walton DM, MacDermid JC. Depression affects the recovery trajectories of patients with distal radius fractures: A latent growth curve analysis. Musculoskelet Sci Pract. 2019 Oct;43:96-102. doi: 10.1016/j.msksp.2019.07.012. Epub 2019 Jul 27. PMID 31374477
- [Background] Scheim AI, Bauer GR. The Intersectional Discrimination Index: Development and validation of measures of self-reported enacted and anticipated discrimination for intercategorical analysis. Soc Sci Med. 2019 Apr;226:225-235. doi: 10.1016/j.socscimed.2018.12.016. Epub 2019 Jan 21. PMID 30674436
- [Background] Shi Q, Sinden K, MacDermid JC, Walton D, Grewal R. A systematic review of prognostic factors for return to work following work-related traumatic hand injury. J Hand Ther. 2014 Jan-Mar;27(1):55-62; quiz 62. doi: 10.1016/j.jht.2013.10.001. Epub 2013 Oct 21. PMID 24268193
- [Background] Walton, D. et al. (2008) 'Prognostic Factors After Acute Whiplash Injury: Results Of A Meta-analysis', Journal of Orthopaedic & Sports Physical, 38(1), p. A23.
- [Background] Walton DM, Carroll LJ, Kasch H, Sterling M, Verhagen AP, Macdermid JC, Gross A, Santaguida PL, Carlesso L; ICON. An Overview of Systematic Reviews on Prognostic Factors in Neck Pain: Results from the International Collaboration on Neck Pain (ICON) Project. Open Orthop J. 2013 Sep 20;7:494-505. doi: 10.2174/1874325001307010494. eCollection 2013. PMID 24115971
- [Background] Walton DM, Krebs D, Moulden D, Wade P, Levesque L, Elliott J, MacDermid JC. The Traumatic Injuries Distress Scale: A New Tool That Quantifies Distress and Has Predictive Validity With Patient-Reported Outcomes. J Orthop Sports Phys Ther. 2016 Oct;46(10):920-928. doi: 10.2519/jospt.2016.6594. Epub 2016 Sep 3. PMID 27594662
- [Background] Walton DM, Mehta S, Seo W, MacDermid JC. Creation and validation of the 4-item BriefPCS-chronic through methodological triangulation. Health Qual Life Outcomes. 2020 May 7;18(1):124. doi: 10.1186/s12955-020-01346-8. PMID 32381020
- [Background] Walton DM, Elliott JM, Lee J, Fakhereddin M, Seo W. Identification of clinically-useful cut scores of the Traumatic Injuries Distress Scale (TIDS) for predicting rate of recovery following musculoskeletal trauma. PLoS One. 2021 Mar 23;16(3):e0248745. doi: 10.1371/journal.pone.0248745. eCollection 2021. PMID 33755664
- [Background] Walton DM, Elliott JM. An Integrated Model of Chronic Whiplash-Associated Disorder. J Orthop Sports Phys Ther. 2017 Jul;47(7):462-471. doi: 10.2519/jospt.2017.7455. Epub 2017 Jun 16. PMID 28622487
- [Background] Walton DM, Elliott JM. A new clinical model for facilitating the development of pattern recognition skills in clinical pain assessment. Musculoskelet Sci Pract. 2018 Aug;36:17-24. doi: 10.1016/j.msksp.2018.03.006. Epub 2018 Apr 9. PMID 29669311
- [Background] Walton DM, Marsh J. Reliability, Discriminative, and Prognostic Validity of the Multidimensional Symptom Index in Musculoskeletal Trauma. Clin J Pain. 2020 Sep;36(9):700-706. doi: 10.1097/AJP.0000000000000856. PMID 32520818
- [Background] Walton DM, Phares P. The potential and perils of prognosticating persistent post-traumatic problems from a postpositivist perspective. Spine J. 2018 Aug;18(8):1483-1488. doi: 10.1016/j.spinee.2018.01.015. Epub 2018 Jan 31. PMID 29355787
- [Background] Walton DM, Beattie T, Putos J, MacDermid JC. A Rasch analysis of the Brief Pain Inventory Interference subscale reveals three dimensions and an age bias. J Clin Epidemiol. 2016 Jun;74:218-26. doi: 10.1016/j.jclinepi.2015.10.022. Epub 2016 Jan 6. PMID 26769256
- [Background] Walton DM, Putos J, Beattie T, MacDermid JC. Confirmatory factor analysis of 2 versions of the Brief Pain Inventory in an ambulatory population indicates that sleep interference should be interpreted separately. Scand J Pain. 2016 Jul;12:110-116. doi: 10.1016/j.sjpain.2016.05.002. Epub 2016 May 25. PMID 28850482
- [Background] Walton DM, Elliott JM, Salim S, Al-Nasri I. A reconceptualization of the pain numeric rating scale: Anchors and clinically important differences. J Hand Ther. 2018 Apr-Jun;31(2):179-183. doi: 10.1016/j.jht.2017.12.008. Epub 2018 Feb 9. No abstract available. PMID 29433765
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235